CLINICAL TRIAL: NCT01169389
Title: Analgesic Control Following Knee Arthroscopy: Results of a Randomised , Double-blinded Trial Comparing a Hyaluronic Acid Supplement to Bupivacaine
Brief Title: Analgesic Control Following Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Research and Innovation Foundation, Ireland (Other)
Responsible Party: Kevin Mulhall, Orthopaedic Research and Innovation Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KM/10/2008/18
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2008-12

CONDITIONS: Knee; Arthroscopy; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Injections, Intra-Articular; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Durolane (Active Comparator)
  Interventions: Procedure: Intraarticular injection
- Bupivacaine (Placebo Comparator)
  Interventions: Procedure: Intra-articular injection of 0.5% Bupivacaine

INTERVENTIONS:
Procedure: Intraarticular injection — Durolane, one vial
  Arms: Durolane
Procedure: Intra-articular injection of 0.5% Bupivacaine
  Arms: Bupivacaine

SUMMARY:
This study aims to investigate the analgesic effects offered by bupivacaine and Durolane (a hyaluronic acid supplement) administered immediately following the completion of knee arthroscopy.

DETAILED DESCRIPTION:
There is increasing evidence of the toxic effects of intraarticular administration of local anaesthetic. Hyaluronic acid supplementation given at the time of knee arthroscopy has not been fully evaluated as a possible alternative. We have studied the efficacy of a hyaluronic acid (HA) supplement (Durolane®) and a local anaesthetic (Bupivacaine) at providing early and short-term post-operative analgesic control following knee arthroscopy.Patients will be randomised to receive either 10mls of 0.5% Bupivacaine or 10mls of Durolane® into the joint immediately after completion of surgery. WOMAC and Tegner-Lysholm scores were obtained at baseline then at 1, 2, and 6-weeks post surgery. VAS pain scores were obtained at baseline; 1 and 24-hours; and 1, 2 and 6 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* those undergoing knee arthroscopy for: diagnostic purposes, removal of loose bodies, articular cartilage debridement or, meniscectomy
* age over 18 years

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) grade ≥3;
* arthroscopic assisted osteotomies;
* a history of two or more prior procedures on the ipsilateral knee;
* post-operative morbidities indirectly linked to the procedure (e.g. anaesthetic complications, DVT or PE);
* systemic steroid requirements;
* previous intra-articular anaesthetic or steroid injection within the last three months;
* intra-articular HA injection within the last nine months;
* intra-articular sepsis within the previous three months;
* prior history of knee arthroplasty, peri-articular fracture, ligamentous instability, inflammatory arthritis or a previous diagnosis of Complex Regional Pain Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale pain score | 1 day
Visual Analogue Scale pain score | 1 week
Visual Analogue Scale pain score | 2 weeks
Visual Analogue Scale pain score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Mulhall, FRCSI, Principal Investigator — Orthopaedic Research and Innovation Foundation, Ireland
Locations (1):
- Sports Surgery Clinic, Dublin, Ireland